CLINICAL TRIAL: NCT02097433
Title: A Phase 1 Open-label Study To Characterize The Pharmacokinetics Of A Single 45 Mg Oral Dose Of Dacomitinib (Pf-00299804) In Healthy Chinese Subjects
Brief Title: Dacomitinib (PF-00299804) Pharmacokinetics In Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: A7471051
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Dacomitinib; PF299804; pharmacokinetics; healthy; Chinese
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dacomitinib (Experimental)
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — A single 45 mg oral dose of Dacomitinib will be administered under fasted conditions to healthy Chinese volunteers

SUMMARY:
As part of the global clinical development program for Dacomitinib, studies are planned in cancer patients in China. An assessment of Dacomitinib pharmacokinetics in Chinese subjects, as required by the Chinese Health Authorities, is therefore warranted.

The single 45 mg oral dose pharmacokinetics of Dacomitinib will be characterized.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics of Dacomitinib in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese volunteers (individuals currently residing in mainland China, who were born in China, and whose parents are both of Chinese descent).
* Healthy male and/or female (of non-childbearing potential) subjects between the ages of 18 and 45 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests).
* Body Mass Index (BMI) of 19.0 to 24.0 kg/m2; and a total body weight should be 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant dermatologic, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Drug dependency, a positive urine drug screen and/or alcohol dependency.
* Use of tobacco- or nicotine- containing products (or a positive urine cotinine test).
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug or biologic within the last 3 months (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication, whichever is longer.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Dacomitinib | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of Dacomitinib | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]of Dacomitinib | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)of Dacomitinib | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
Apparent Volume of Distribution (Vz/F)of Dacomitinib | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2)of Dacomitinib | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F)of Dacomitinib | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05199265 | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of PF-05199265 | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)of PF-05199265 | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]of PF-05199265 | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Plasma Decay Half-Life (t1/2)of PF-05199265 | predose, 1, 2 ,4, 6, 8, 12, 24, 48 ,72 ,96, 120, 144, 168, 192, 216, 240 ,264 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471051&StudyName=Dacomitinib%20%28PF-00299804%29%20Pharmacokinetics%20In%20Chinese%20Healthy%20Volunteers